CLINICAL TRIAL: NCT04714307
Title: Neuropsychiatry and Cognition in the Context of Spinocerebellar Ataxia Type 3/Machado-Joseph Disease (SCA3/MJD)
Brief Title: Neuropsychiatry and Cognition in SCA3/MJD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: 20190606
Record Dates: First submitted 2020-12-08; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Spinocerebellar Ataxia Type 3; Machado-Joseph Disease; SCA3; MJD
MeSH Terms: conditions — Machado-Joseph Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will be retained under codification for the use of this research only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Symptomatic: Molecularly diagnosed SCA3/MJD Symptomatic subjects.
  Interventions: Diagnostic Test: Cognitive Testing; Diagnostic Test: Psychiatric Evaluation; Diagnostic Test: Clinical Neurological Evaluation; Diagnostic Test: Emotional Attribution Evaluation; Diagnostic Test: Activities of Daily Living
- Non-related Controls: Controls matched with symptomatic by age and educational level.
  Interventions: Diagnostic Test: Cognitive Testing; Diagnostic Test: Psychiatric Evaluation; Diagnostic Test: Emotional Attribution Evaluation
- At 50% risk for SCA3/MJD group: The offspring of affected individuals with SARA<3. This group will be comprised of two subpopulations: pre-symptomatic individuals and related controls. The determination will be made upon molecular diagnosis to be done in a double-blind manner.
  Interventions: Diagnostic Test: SCA3/MJD molecular diagnosis; Diagnostic Test: Cognitive Testing; Diagnostic Test: Psychiatric Evaluation; Diagnostic Test: Clinical Neurological Evaluation; Diagnostic Test: Emotional Attribution Evaluation; Diagnostic Test: Activities of Daily Living

INTERVENTIONS:
Diagnostic Test: SCA3/MJD molecular diagnosis — Double-blind molecular diagnosis for determination of the presence of the mutation.
  Groups: At 50% risk for SCA3/MJD group
Diagnostic Test: Cognitive Testing — Cross-sectional Cognitive evaluation with
  * CCAS Scale
  * Trail-Making Test parts A and B
  * Stroop Color-Word Test
Diagnostic Test: Psychiatric Evaluation — Cross-sectional Psychiatric evaluation with Hamilton-Anxiety and Hamilton-Depression rating scales.
Diagnostic Test: Clinical Neurological Evaluation — Cross-sectional neurological evaluation with standardized clinical scales - SARA, SCAFI and CCFS.
  Groups: At 50% risk for SCA3/MJD group; Symptomatic
Diagnostic Test: Emotional Attribution Evaluation — Cross-sectional emotional attribution evaluation by means of the Reading the Mind in the Eyes Test (RMET).
Diagnostic Test: Activities of Daily Living — Cross-sectional evaluation of Activities of Daily Living (ADLs) by means of Friedreich Ataxia Rating Scale Part II.
  Groups: At 50% risk for SCA3/MJD group; Symptomatic

SUMMARY:
This research investigates how cognitive-affective aspects evolve during the course of SCA3/MJD. Due to COVID-19 pandemics, this study protocol was adapted for online-only consultations. Evaluations happening after March 2020 have been done by videocall with patients, and no neurological evaluation was thus performed on these patients. A scale on Activities of Daily Living was added to the online protocol to replace SARA, SCAFI and CCFS scales.

DETAILED DESCRIPTION:
By the end of this study, the evaluated population will be composed of 144 participants: 36 ataxic SCA3/MJD carriers, 72 at 50% risk of carrying the SCA3/MJD mutation and 36 healthy controls. Ataxic subjects are invited to participate if they have an established molecular diagnosis of SCA3/MJD and have a SARA score greater than 2.5 points. At risk subjects are composed by the offspring of molecularly diagnosed SCA3/MJD subjects that have a SARA<3. Healthy controls belonging either to families living with the disease or to the general population are invited to participate according to how well they match with ataxic subjects included in the study. Subjects are invited to participate in the study and, after constentment procedures, cognitive-affective assessments and a scale on Activities of Daily Living (ADL) are performed on a videocall. At risk subjects collect a blood sample for double bilnd determination of their carrier status. Before March 2020, all procedures were performed in person and, instead of ADL, SARA, SCAFI and CCFS were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic:
* older than 18 year old;
* molecular diagnosis of SCA3/MJD;
* SARA>2.5.
* At 50% risk:
* older than 18 year old;
* have a parent with molecular diagnosis of SCA3/MJD;
* SARA<3.
* Healthy Controls
* older than 18 year old;
* no genetic relationship with a SCA3/MJD carrier.

Exclusion Criteria:

* Non agreement in signing the informed consent;
* Healthy Controls: having any history of genetic disorders in their families or any psychiatric or neurologic disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with molecular diagnosis of SCA3/MJD will be recruited from the Medical Genetics Service database of Hospital de Clínicas de Porto Alegre, Brazil, by telephone calls or by invitation in the outpatient clinic. First degree relatives of these subjects at 50% risk of carrying the mutation will also be invited to participate. Healthy controls will be invited from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Cerebellar Cognitive Affective Syndrome Scale | Through study completion, an average of 1 year
  Study the performance on the Cerebellar Cognitive Affective Syndrome Scale of SCA3/MJD symptomatic subjects when compared to matched healthy controls and of pre-symptomatic subjects when compared to familial healthy controls.
Trail-Making Test Part A and B | Through study completion, an average of 1 year
  Study the performance on the Trail-Making Test Part A and B of SCA3/MJD symptomatic subjects when compared to matched healthy controls and of pre-symptomatic subjects when compared to familial healthy controls.
Stroop Color-Word Test | Through study completion, an average of 1 year
  Study the performance on the Stroop Color-Word Test of SCA3/MJD symptomatic subjects when compared to matched healthy controls and of pre-symptomatic subjects when compared to familial healthy controls.
Emotion Attribution impairment in SCA3/MJD | Through study completion, an average of 1 year
  Study the performance of symptomatic SCA3/MJD carriers in the Reading the Mind in the Eyes Test.
Emotion Attribution in different phases of the disease | Through study completion, an average of 1 year
  Study the performance of pre-symptomatic SCA3/MJD carriers in the Reading the Mind in the Eyes Test.
Hamilton Anxiety Rating Scale | Through study completion, an average of 1 year
  Study the profile of symptomatic and pre-symptomatic SCA3/MJD carriers in the Hamilton Anxiety Rating Scale.
Hamilton Depression Rating Scale | Through study completion, an average of 1 year
  Study the profile of symptomatic and pre-symptomatic SCA3/MJD carriers in the Hamilton Depression Rating Scale.

SECONDARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia (SARA) | Through study completion, an average of 1 year
  Correlations between primary outcomes and SARA.
Composite Cerebellar Functional Severity Score (CCFS) | Through study completion, an average of 1 year
  Correlations between primary outcomes and CCFS.
SCA Functional Index | Through study completion, an average of 1 year
  Correlations between primary outcomes and SCAFI.
Friedreich Ataxia Rating Scale part II (FARS part II) | Through study completion, an average of 1 year
  Correlations between primary outcomes and Activities of Daily Living from FARS part II.

CONTACTS AND LOCATIONS:
Overall Officials: Laura B. Jardim, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre and Universidade Federal do Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be done via direct contact with the Principal Investigator in order to preserve individual participants identities.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will become available after final statistical analysis and data publishing via direct contact with principal investigator.
Access Criteria: Investigators and researchers of the area